CLINICAL TRIAL: NCT02947165
Title: A Phase I/Ib, Open-label, Multi-center Dose Escalation Study of NIS793 in Combination With PDR001 in Adult Patients With Advanced Malignancies
Brief Title: Phase I/Ib Study of NIS793 in Combination With PDR001 in Patients With Advanced Malignancies.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNIS793X2101; 2016-003044-36 (EudraCT Number)
Record Dates: First submitted 2016-10-18; First posted 2016-10-27 (Estimated); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer; Lung Cancer; Hepatocellular Cancer; Colorectal Cancer; Pancreatic Cancer; Renal Cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Liver Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Kidney Neoplasms | interventions — NIS-793; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NIS793 (Experimental)
  Interventions: Drug: NIS793
- NIS793 + PDR001 (Experimental)
  Interventions: Drug: NIS793; Drug: PDR001

INTERVENTIONS:
Drug: NIS793 — Anti-TGF beta antibody tested on a Q3W regimen or alternative Q2W regimen.
Drug: PDR001 — Anti-PD-1 antibody tested on a Q3W regimen or alternative Q4W regimen.
  Arms: NIS793 + PDR001

SUMMARY:
To characterize the safety and tolerability of NIS793 as single agent and in combination with PDR001 and to identify recommended doses for future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained prior to any screening procedures.
2. Patient (male or female) ≥ 18 years of age.
3. Escalation: Patients with advanced/metastatic solid tumors, with measurable or non-measurable disease as determined by RECIST version 1.1 who have progressed despite standard therapy or are intolerant of standard therapy, or for whom no standard therapy exists.
4. Expansion: Patients with advanced/metastatic solid tumors, with at least one measurable lesion as determined by RECIST version 1.1, who have progressed despite standard therapy following their last prior therapy or are intolerant to standard therapy and fit into one of the following groups: Group 1: NSCLC resistant to anti-PD-1/PD-L1; Group 2: TNBC; Group 3: HCC; Group 4: MSS-CRC; Group 5: pancreatic; Group 6 ccRCC resistant to anti-PD-1/PD-L1.

   Resistance to anti-PD-1/PD-L1 therapy is defined as: Documented progressive disease occurring while on/or within 6 months after anti-PD-1 and/or anti-PD-L1 agent (single or combination) received as the last therapy prior to enrollment.
5. ECOG Performance Status ≤ 2.
6. Patients must have a site of disease amenable to biopsy, and be a candidate for tumor biopsy. Patient must be willing to undergo a new tumor biopsy at screening, and during therapy on this study. Exceptions may be made on a case by case basis after documented discussion with Novartis.

Exclusion Criteria:

1. History of severe hypersensitivity reactions to study treatment ingredients or other monoclonal antibodies and components of study drug.
2. Patients with active, known or suspected autoimmune disease. Note: Patients with vitiligo, type I diabetes mellitus, residual hypothyroidism only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
3. HIV infection.
4. Active HBV or HCV infection.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Incidence of DLTs, AEs, SAEs and dose reductions / interruptions for NIS793 | Up to 90 days after end of treatment
Incidence of DLTs, AEs, SAEs and dose reductions/interruptions for NIS793 in combination with PDR001 | Up to 150 days after end of treatment

SECONDARY OUTCOMES:
Best overall response (BOR) | 48 months
  Evaluate the anti-tumor activity per RECIST as well as per immune related Response Criteria (irRC) of NIS793 as single agent and in combination with PDR001 every 2 cycles from start of treatment until cycle 9 then every 3 cycles until end of treatment (if applicable).
Disease control rate (DCR) | 48 months
  Evaluate the anti-tumor activity per RECIST as well as per immune related Response Criteria (irRC) of NIS793 as single agent and in combination with PDR001every 2 cycles from start of treatment until cycle 9 then every 3 cycles until end of treatment (if applicable).
Overall response rate (ORR) | 48 months
  Evaluate the anti-tumor activity per RECIST as well as per immune related Response Criteria (irRC) of NIS793 as single agent and in combination with PDR001 every2 cycles from start of treatment until cycle 9 then every 3 cycles until end of treatment (if applicable).
Progression free survival (PFS) | 48 months
  Evaluate the anti-tumor activity per RECIST as well as per immune related Response Criteria (irRC) of NIS793 as single agent and in combination with PDR001 every 2 cycles from start of treatment until cycle 9 then every 3 cycles until end of treatment. During disease progression f/u, every 8 weeks for 40 weeks, then every 12 weeks.
Duration of response (DOR) | 48 months
  Evaluate the anti-tumor activity per RECIST as well as per immune related Response Criteria (irRC) of NIS793 as single agent and in combination with PDR001 every 2 cycles from start of treatment until cycle 9 then every 3 cycles until end of treatment (if applicable).
Serum concentration-time profiles of NIS793 single agent and NIS793 in combination with PDR001 | 48 months
  Evaluate serum concentration of NIS793 and PDR001 up to 8 cycles after start of treatment and at end of treatment.
Presence of anti-NIS793 and anti-PDR001 antibodies | 48 months
  Assess the emergence of anti-NIS793 and anti-PDR001 antibodies up to 8 cycles after start of treatment and at end of treatment.
Concentration of anti-NIS793 and anti-PDR001 antibodies | 48 months
  Assess the concentration of anti-NIS793 and anti-PDR001 antibodies up to 8 cycles after start of treatment and at end of treatment.
Area under the curve (AUC) for NIS793 single agent and NIS793 in combination with PDR001. | 48 months
  Characterize the pharmacokinetic properties of NIS793 given alone and in combination with PDR001.
Cmax for NIS793 single agent and NIS793 in combination with PDR001. | 48 months
  Characterize the pharmacokinetic properties of NIS793 given alone and in combination with PDR001.
Tmax for NIS793 single agent and NIS793 in combination with PDR001. | 48 months
  Characterize the pharmacokinetic properties of NIS793 given alone and in combination with PDR001.
Half life of NIS793 as single agent and in combination with PDR001. | 48 months
  Characterize the pharmacokinetic properties of NIS793 given alone and in combination with PDR001.
Characterization of tumor infiltrating lymphocytes (TILs) by H&E | 48 months
  Assess change from baseline of immune infiltrates in tumor biopsies after 2 cycles of treatment.
Characterization of tumor infiltrating lymphocytes by immunohistochemistry using markers such as CD8 and PD-L1 | 48 months
  Assess change from baseline in immunological markers in tumor biopsies after 2 cycles of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (2):
  - Sarah Cannon Research Institute SC, Nashville, Tennessee
  - Huntsman Cancer Institute SC, Salt Lake City, Utah
- Novartis Investigative Site, Salzburg, Austria
- Novartis Investigative Site, Toronto, Ontario, Canada
- Germany (2):
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Hong Kong, Hong Kong
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
- Novartis Investigative Site, Kashiwa, Chiba, Japan
- Novartis Investigative Site, Sankt Gallen, Switzerland
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bauer TM, Santoro A, Lin CC, Garrido-Laguna I, Joerger M, Greil R, Spreafico A, Yau T, Goebeler ME, Hutter-Kronke ML, Perotti A, Juif PE, Lu D, Barys L, Cremasco V, Pelletier M, Evans H, Fabre C, Doi T. Phase I/Ib, open-label, multicenter, dose-escalation study of the anti-TGF-beta monoclonal antibody, NIS793, in combination with spartalizumab in adult patients with advanced tumors. J Immunother Cancer. 2023 Nov 29;11(11):e007353. doi: 10.1136/jitc-2023-007353. PMID 38030303
- [Derived] Dodagatta-Marri E, Meyer DS, Reeves MQ, Paniagua R, To MD, Binnewies M, Broz ML, Mori H, Wu D, Adoumie M, Del Rosario R, Li O, Buchmann T, Liang B, Malato J, Arce Vargus F, Sheppard D, Hann BC, Mirza A, Quezada SA, Rosenblum MD, Krummel MF, Balmain A, Akhurst RJ. alpha-PD-1 therapy elevates Treg/Th balance and increases tumor cell pSmad3 that are both targeted by alpha-TGFbeta antibody to promote durable rejection and immunity in squamous cell carcinomas. J Immunother Cancer. 2019 Mar 4;7(1):62. doi: 10.1186/s40425-018-0493-9. PMID 30832732